CLINICAL TRIAL: NCT02643147
Title: Loop Diuretic Dosage in Patients With Acute Heart Failure and Renal Failure: Conventional Versus Carbohydrate Antigen 125-guided Therapy (IMPROVE-HF)
Acronym: IMPROVE-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Julio Nuñez, MD, PhD, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-001433-83
Record Dates: First submitted 2015-12-14; First posted 2015-12-31 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Renal Failure; Biomarker guided-therapy; Loop diuretics; Carbohydrate antigen 125
MeSH Terms: conditions — Heart Failure; Renal Insufficiency | interventions — Sodium Potassium Chloride Symporter Inhibitors; Furosemide; CA-125 Antigen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CA125 guided strategy (Experimental): In this group loop diuretic (Furosemide) dosage will be guided by Carbohydrate Antigen 125 (CA125) plasma levels
  Interventions: Drug: CA125 guided strategy
- Conventional strategy (Active Comparator): Standard treatment strategy Therapy is based on established european guidelines
  Interventions: Drug: Conventional Strategy

INTERVENTIONS:
Drug: CA125 guided strategy — Initial dose of intravenous furosemide ≤80 mg / day regardless of prior dose of loop diuretics who were receiving.
  Other Names: Loop diuretic (Furosemide) dosage in CA125 ≤35 U/ml patients
  Arms: CA125 guided strategy
Drug: CA125 guided strategy — Initial dose of intravenous furosemide ≥120 mg/day or 2.5 times the dose the patient was taking at home.
  Other Names: Loop diuretic dosage (Furosemide) in CA125 >35 U/ml patients
  Arms: CA125 guided strategy
Drug: Conventional Strategy — The dosage of loop diuretics is done according to the presence of symptoms and signs of systemic congestion and current recommendations
  Arms: Conventional strategy

SUMMARY:
Worsening renal function (WRF) is a frequent finding in patients with decompensated acute heart failure (AHF) and it is associated to increased length of hospitalization and higher morbidity and mortality. Traditionally, WRF in AHF setting has been attributed to low cardiac output, but recent evidence also suggests venous congestion play a crucial role. Loop diuretics are the mainstay treatment of AHF, but their use traditionally has been associated to WRF, but also renal function improvement in patients with unequivocal signs of congestion. Nevertheless, traditional symptoms or signs of patients with AHF have shown a limited accuracy to neither identify nor quantify the degree of venous congestion. Recent authors have reported that plasma levels of antigen carbohydrate 125 (CA125) are closely related to the degree of venous congestion.

The investigators hypothesize that CA125 may have a role for identifying the hyperhydrated (High CA125) patients that need high loop diuretic doses, and those with normal CA125 values needing low loop diuretic doses. In this randomized study (1:1) the investigators seek to evaluate whether a CA125 loop diuretic guided management therapy is superior to a standard strategy. The primary endpoint is the magnitude of changes of renal function at 24 and 72 hours after initiation of intravenous diuretic in an acute worsening of heart failure

ELIGIBILITY:
Inclusion Criteria:

Patients with the diagnosis of acute heart failure (AHF) and the concurrence of the following conditions:

1. Presence of symptoms (dyspnea at rest or minimal exertion) and signs attributable to congestion (signs of congestion on chest radiography, or presence of peripheral edema or ascites, or jugular venous distension at 45 degrees or presence of crackles on auscultation).
2. Elevated natriuretic peptide (NT-proBNP> 1000 pg/ml or BNP> 100 mg/dl).
3. Creatinine ≥1,4 mg/dl on admission, provided that the estimated glomerular filtration rate less than 60 ml / min / m2.
4. Intent to be treated with loop diuretics intravenously.

Exclusion Criteria:

1. Life expectancy less than 6 months of life due to other comorbid conditions.
2. Cardiogenic shock.
3. Diagnosis of acute coronary syndrome in the previous 30 days.
4. Pregnancy at the time of inclusion.
5. Restrictive or Obstructive pulmonary disease or severe degree.
6. Chronic renal insufficiency in stage V (estimated glomerular filtration rate <15 ml / min / m2) or patient previously included in known dialysis program.
7. Participation in another clinical trial randomized at the time of inclusion.
8. Temperature ≥38 ° C or diagnosis of pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Change in renal function (GFR) | 24 and 72 hours
  Glomerular filtration rate (GFR) estimated by MDRD. Prespecified interim analysis of primary outcome will be made by protocol when first 100 patients are included.

SECONDARY OUTCOMES:
Improvement in signs and symptoms of heart failure (NYHA) | 24 and 72 hours
  Evaluation of dyspnea (changes in the functional class of the New York Heart Association -NYHA)
Improvement in signs and symptoms of heart failure (VAS) | 24 and 72 hours
  Evaluation of signs of systemic congestion, and patient global assessment (by visual analogue scale -VAS-)
Changes in plasma levels of natriuretic peptide (NT-proBNP) | 72 hours
Changes in plasma levels of high sensitive troponin | 72 hours
Time required to change intravenous diuretics to oral administration. | Through study completion (30-day follow-up)
Composite of all-cause mortality plus acute heart failure related rehospitalization | 30 days
  Number of events in each group during 30-day follow-up
Change in renal function (creatinin) | 24 h, 72 h and 30 days
  Serum levels of creatinine
Change in renal function (urea) | 24 h, 72 h and 30 days
  Serum levels of urea
Change in renal function (cystatin C) | 24 h, 72 h and 30 days
  Serum levels of Cystatin C

CONTACTS AND LOCATIONS:
Overall Officials: Julio Nuñez, MD, PhD, Principal Investigator — Fundación para la Investigación del Hospital Clínico de Valencia
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain

REFERENCES:
- [Derived] de la Espriella R, Nunez E, Llacer P, Garcia-Blas S, Ventura S, Nunez JM, Sanchez R, Facila L, Vaquer JM, Bodi V, Santas E, Minana G, Mollar A, Nunez G, Chorro FJ, Gorriz JL, Sanchis J, Bayes-Genis A, Nunez J. Early urinary sodium trajectory and risk of adverse outcomes in acute heart failure and renal dysfunction. Rev Esp Cardiol (Engl Ed). 2021 Jul;74(7):616-623. doi: 10.1016/j.rec.2020.06.004. Epub 2020 Jul 2. English, Spanish. PMID 32624444